CLINICAL TRIAL: NCT06929000
Title: A Study on Application of Adjustable Headrest in Painless Curettage Surgery for Overweight and Obese Patients: a Randomized Controlled Trial
Brief Title: A Study on Application of Adjustable Headrest in Painless Curettage Surgery for Overweight and Obese Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCHH_010
Record Dates: First submitted 2025-03-27; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Adjustable Headrests; Ventilation Function; Obese Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the adjustable headrest group: placing an adjustable pillows on the head (Experimental): the adjustable headrest group: placing an adjustable pillows on the patient's head to align the patient's external auditory canal horizontally with the sternum
  Interventions: Other: the adjustable headrest group
- the supine head-lateral position group (Active Comparator): the supine head-lateral position group: during the perioperative period, keep the patient's head tilted to the left or right
  Interventions: Other: the supine head-lateral position group
- the supine head-straight position group (Placebo Comparator): the supine head-straight position group: during the perioperative period, keep the patient's head upright
  Interventions: Other: the supine head-straight position group

INTERVENTIONS:
Other: the supine head-lateral position group — the supine head-lateral position group: during the perioperative period, keep the patient's head tilted to the left or right
  Arms: the supine head-lateral position group
Other: the adjustable headrest group — the adjustable headrest group: placing an adjustable pillows on the patient's head to align the patient's external auditory canal horizontally with the sternum
  Arms: the adjustable headrest group: placing an adjustable pillows on the head
Other: the supine head-straight position group — the supine head-straight position group: during the perioperative period, keep the patient's head upright
  Arms: the supine head-straight position group

SUMMARY:
The aim of this study is to observe the effect of adjustable headrests on ventilation function in overweight and obese patients through clinical experiments, and to explore the impact on the incidence of hypoxemia during painless curettage in overweight and obese patients.

Participants will be randomly allocated to three groups: the supine head-straight position group(Group A), the supine head-lateral position group(Group B), and the adjustable headrest group(Group C). These three groups of patients underwent painless curettage surgery in the daytime operating room and the occurrence of hypoxemia will be observed.

ELIGIBILITY:
Inclusion Criteria:

* patients who choose to have painless surgical abortion
* Body mass index greater than 24
* the American Society of Anesthesiologists (ASA) physical status ranked I-II
* competent to provide informed consent

Exclusion Criteria:

* Abnormal lung function or respiratory system diseases
* Airway obstruction or respiratory malformation
* cervical spondylosis
* psychiatric disorders

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia | 1,2 and 3 minutes after anesthesia induction
  Incidence of hypoxemia will be recorded after anesthesia induction
Respiratory rate and oxygen saturation | The time of entering the daytime operating room, intraoperative period., 1 minute after the patient wakes up
  Respiratory rate and oxygen saturation will be recorded at 4 time points, including the time of entering the daytime operating room(Time 0), 1 minute after anesthesia induction(Time 1), 2 minute after anesthesia induction(Time 2), 3 minute after anesthesia induction(Time 3), 1 minute after the patient wakes up(Time 4)

SECONDARY OUTCOMES:
Heart rate and blood pressure | The time of entering the daytime operating room, intraoperative period, 1 minute after the patient wakes up
  heart rate and blood pressure will be recorded at 4 time points, including the time of entering the daytime operating room(Time 0), 1 minute after anesthesia induction(Time 1), 2 minute after anesthesia induction(Time 2), 3 minute after anesthesia induction(Time 3), 1 minute after the patient wakes up(Time 4)

CONTACTS AND LOCATIONS:
Overall Officials: Na Li NaLi, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes